CLINICAL TRIAL: NCT02328313
Title: LCCC 1410: Impact of Physical Activity on Biomarker of Aging and Body Composition Among Breast Cancer Survivors Age 65 and Older
Brief Title: Impact of Physical Activity on Biomarker of Aging and Body Composition Among Breast Cancer Survivors Age 65 and Older
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LCCC1410; 14-2074 (Other: UNC IRB)
Record Dates: First submitted 2014-10-21; First posted 2014-12-31 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer; Aging; Physical Activity
Keywords: Cancer; Breast Cancer; Geriatric; Advance Age; Exercise; Physical Activity; Genetic Marker; p16; Chemotherapy; Breast Cancer Treatment
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Neoplasms | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention Cohort (Experimental): Breast cancer patients 65 and older undergoing chemotherapy and participating in a home-based physical activity intervention.
  Interventions: Behavioral: Walk with Ease Program

INTERVENTIONS:
Behavioral: Walk with Ease Program — The Walk With Ease Program sets a goal for participants to walk 30 minutes a day five times a week and gives helpful hints on how to achieve this goal.

SUMMARY:
To determine if exercise will affect the increase in p16 expression that is associated with both chemotherapy administration and advancing age.

DETAILED DESCRIPTION:
LCCC1410 is designed to compare the change in p16 from baseline to end of chemotherapy in 100 older (≥ 65 years) breast cancer patients participating in a home-based physical activity program (intervention group) to 100 patients in the concurrent control group not participating in a physical activity intervention (enrolled in a separate RO1 study as described in section 1.7). The biomarker p16 is known to dramatically increase with chemotherapy, and we hypothesize that the increase will be attenuated by a physical activity intervention. We will evaluate changes in p16 between the two study populations. Data from the geriatric assessment at baseline will be used to characterize the study population, and subscale scores from the GA will also be assessed for differences between baseline and end of chemotherapy to compare the LCCC1410 study population with the concurrent control.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older, female
* Histologically confirmed Stage I, II or III breast cancer (if the patient has had more than one breast cancer, then the most recent diagnosis)
* Scheduled to begin an appropriate adjuvant or neoadjuvant chemotherapy regimen as defined by NCCN guidelines (www.nccn.org)
* English speaking
* IRB approved, signed written informed consent
* Approval from their treating physician to engage in moderate-intensity physical activity
* Patient-assessed ability to walk and engage in moderate physical activity
* Willing and able to meet all study requirements.

Exclusion Criteria:

- One or more significant medical conditions that in the physician's judgment preclude participation in the walking intervention.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-10; Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
To measure the change in level of p16 expression from baseline to end of chemotherapy to a control group | 12 months
  The comparison group will be taken from another study
To measure the changes in the level of p16 expression from baseline and end of chemotherapy. | 2 - 6 months
  The study will look at the change of p16 expression within patients on this study.

SECONDARY OUTCOMES:
To measure changes in body compositional aspects of lean body mass (LBM) | 12 months
  As measured by DEXA
To measure changes in body compositional aspects of fat tissue mass (FM) | 12 months
  As measured by DEXA
To measure changes in body compositional aspects of percentage body fat (BF) | 12 months
  As measured by DEXA
To measure change in physical activity over the course of the study | 12 months
  As measured by engagement in walking survey
To measure change in physical function over the course of the study | 12 months
  As measured by the Short Physical Performance Battery
To measure change in fatigue over the course of the study | 12 months
  As measured by the FACIT-F
To measure change in quality of life over the course of the study | 12 months
  As measured by the FACT-B
To measure change in self-efficacy over the course of the study | 12 months
  As measured by the PSEFSM and OEE
To measure retention during the study | 12 months
  • Retention will be assessed as the proportion of patients who enroll in the study who complete all questionnaires and assessments at all time points.
To measure safety of the walking program | 12 months
  • Safety will be defined as any adverse events potentially related to the intervention, including falls, which are reported by study participants to the Study Team.
To measure overall satisfaction with the program | 12 months
  As measured by a satisfaction questionnaire
To average the number of daily and weekly steps per participant | 12 months
  As measure via an continuous accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Hyman Muss, MD, Principal Investigator — University of North Carolina
Locations (1):
- Amy Garrett, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Nyrop KA, Page A, Deal AM, Wagoner C, Kelly EA, Kimmick GG, Copeland A, Speca J, Wood WA, Muss HB. Association of self-directed walking with toxicity moderation during chemotherapy for the treatment of early breast cancer. Support Care Cancer. 2023 Dec 28;32(1):68. doi: 10.1007/s00520-023-08275-4. PMID 38153568